CLINICAL TRIAL: NCT03855046
Title: A Comparative Efficacy and Safety Study of Lateral Subcutaneous Sphincterotomy and Botulinum Toxin Type A in the Treatment of Chronic Anal Fissure
Brief Title: Complex Treatment of a Chronic Anal Fissure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Collaborators: St. Petersburg State Pavlov Medical University (Other); Astrakhan State Medical University (Other); Siberian State Medical University (Other); City Clinical Hospital №24, Department of Health City of Moscow (Other Government); GBUZ MO "Lvovskaia Raionaia Bolnica" (Other Government); Medical Center ON-CLINIC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56IG701SSCC978
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Fissure in Ano
Keywords: Internal sphincterotomy; Anal fissure; Chronic anal fissure; botulinum toxin A; proctologic diseases; surgical treatment; Chronic anal pain; Fecal incontinence; Spasm of the internal sphincter; Anal sphincter insufficiency; randomized
MeSH Terms: conditions — Fissure in Ano; Fecal Incontinence | interventions — incobotulinumtoxinA; Solutions

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, randomized, controlled clinical study. Surgical removal of anal fissure followed by internal sphincter relaxation with Botulinum toxin type A is performed in the study group.
  Lateral subcutaneous sphincterotomy to relax sphincter is a method of choice in the control group. Patients are randomized with envelope method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xeomin (Experimental): Complex treatment of chronic anal fissure with drug-induced relaxation of the internal sphincter with Botulinum Toxin Type A. (IncobotulinumtoxinA 50 U Intramuscular Powder for Solution).
  Interventions: Drug: IncobotulinumtoxinA 50 U Intramuscular Powder for Solution
- Xeomin control (Active Comparator): Complex treatment of chronic anal fissure with lateral subcutaneous sphincterotomy.
  Interventions: Procedure: Lateral subcutaneous sphincterotomy.

INTERVENTIONS:
Drug: IncobotulinumtoxinA 50 U Intramuscular Powder for Solution — Sparing surgical removal of fissure without internal sphincter incision is held under spinal anesthesia in surgical room at lithotomy position using electrocoagulation.
  After that Botulinum Toxin Type A is injected into the internal anal sphincter at 1, 5, 7 and 11 o'clock (localization of injection points), 10 U at each point (40 U in total). Botulinum toxin type A (a 50 U vial) is diluted with 1.0 ml of 0.9% saline solution.
  Other Names: Xeomin
  Arms: Xeomin
Procedure: Lateral subcutaneous sphincterotomy. — The patient is positioned on the table like for perineal lithotomy. After spinal anesthesia, the anal canal and then the surgical field are treated with 70% ethanol. Under the rectal speculum control, sparing surgical removal of fissure without internal sphincter incision is held using electrocoagulation.Then, in a 3 or 9 o'clock position, a narrow (eye) scalpel is inserted into the intersphincteric groove separating the external and internal sphincters, the scalpel blade is turned to the rectal lumen, and the internal sphincter is dissected up to the wall of the anal canal mucosa under the control of the finger inserted into the anal canal. After controlling hemostasis, the operation is ended with the introduction of the vent tube and hemostatic sponge.
  Arms: Xeomin control

SUMMARY:
This study is aimed at studying the efficacy and safety of treating chronic anal fissure with botulinum toxin versus lateral subcutaneous sphincterotomy.

DETAILED DESCRIPTION:
Chronic anal fissure is a rupture of anal canal mucosa lasting for more than 2 months and resistant to non-surgical treatment. This condition is attended by severe pain syndrome during and after bowel movement (defecation). This condition is most frequent in younger and working-age adults; therefore, the treatment issue is of particular relevance.

The main cause of chronic anal fissure development is spasm of the internal sphincter. It should be eliminated in the first instance, in order to provide the effective therapy. All the main treatment methods, such as medicinal relaxation of the internal sphincter with 0.4% nitroglycerin ointment, lateral subcutaneous sphincterotomy, and pneumodivulsion of the anal sphincter are aimed at its removal. However, the optimal method has not yet been developed.

Non-surgical treatments are often attended by relapse of disease, while surgical treatment is often complicated by intestinal contents incontinence, usually gas and loose or hard stool in some occasions (grade 3 anal sphincter insufficiency).

In particular, lateral subcutaneous sphincterotomy performed in such patients is associated with an increase in the degree of anal incontinence in the early post-operative period.

Botulinum Toxin Type A application in complex treatment of patients with chronic anal fissure (after fissure excision) is intended to improve the therapy results, namely to reduce the frequency and duration of anal sphincter insufficiency after sphincter spasm removal (reduction in the number of patients suffering from post-operative incontinence).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic anal fissure

Exclusion Criteria:

* Inflammatory diseases of the colon
* Pectenosis
* Previous surgical interventions on the anal canal
* IV grade internal and external hemorrhoids
* Rectal fistula
* Severe somatic diseases at the decompensation stage
* Pregnancy and lactation
* Individual intolerance and hypersensitivity to botulinum toxin
* Myasthenia gravis and myasthenia-like syndromes
* Anal sphincter insufficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Anal sphincter insufficiency | Up to 60 days
  Frequency of anal sphincter insufficiency according to the Wexner scale incontinence after the surgical intervention. Self reported daily meausure outcome, wich evaluate from 0 - to 20 points (where 0 points = full feacal continence; 20 points = full feacal incontinence).

SECONDARY OUTCOMES:
2-item pain intensity (P2) | On day 7, 30 and 60
  Self reported pain intensity after the defecation and during the day after the surgical intervention. Each item is scored 0-10 (0 = no pain; 10 = pain as bad, as can can be).
Non-Healing Wound | On day 60
  Frequency of post-operative wound epithelialization
Profilometry /sphincterometry findings | On day 30 and 60
  Internal sphincter spasm or local internal sphincter spasm by the data of anorectal profilometry / or anorectal sphincterometry
Temporary disability | Up to 60 days
  Duration of temporary disability
Relap | Up to 60 days
  Frequency of relapses

CONTACTS AND LOCATIONS:
Overall Officials: Sergey A. Frolov, Ph.D., Principal Investigator — State Scientific Centre of Coloproctology, Russian Federation (SSCCRussia)
Locations (7):
- Russia (7):
  - GBUZ MO "Lvovskaia Raionaia Bolnica", Podolsk, Moscow Oblast
  - Astrakhan State Medical University, Astrakhan
  - Medical Center ON-CLINIC, Moscow
  - SSCCRussia, Moscow
  - City Clinical Hospital №24, Department of Health City of Moscow, Moscow
  - St. Petersburg State Pavlov Medical University, Saint Petersburg
  - Siberian State Medical University, Tomsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart DB Sr, Gaertner W, Glasgow S, Migaly J, Feingold D, Steele SR. Clinical Practice Guideline for the Management of Anal Fissures. Dis Colon Rectum. 2017 Jan;60(1):7-14. doi: 10.1097/DCR.0000000000000735. No abstract available. PMID 27926552
- [Background] Sohn N, Eisenberg MM, Weinstein MA, Lugo RN, Ader J. Precise anorectal sphincter dilatation--its role in the therapy of anal fissures. Dis Colon Rectum. 1992 Apr;35(4):322-7. doi: 10.1007/BF02048108. PMID 1582352
- [Background] Renzi A, Izzo D, Di Sarno G, Talento P, Torelli F, Izzo G, Di Martino N. Clinical, manometric, and ultrasonographic results of pneumatic balloon dilatation vs. lateral internal sphincterotomy for chronic anal fissure: a prospective, randomized, controlled trial. Dis Colon Rectum. 2008 Jan;51(1):121-7. doi: 10.1007/s10350-007-9162-7. Epub 2007 Dec 15. PMID 18080713
- [Background] Gui D, Cassetta E, Anastasio G, Bentivoglio AR, Maria G, Albanese A. Botulinum toxin for chronic anal fissure. Lancet. 1994 Oct 22;344(8930):1127-8. doi: 10.1016/s0140-6736(94)90633-5. PMID 7934496
- [Background] Khan M.I., Khan H., Khan A.U., et. al. Comparing the efficacy of botulinum toxin injection and lateral internal sphincterotomy for chronic anal fissure. KJMS, 2016. 9(1): p. 6
- [Background] Bobkiewicz A, Francuzik W, Krokowicz L, Studniarek A, Ledwosinski W, Paszkowski J, Drews M, Banasiewicz T. Botulinum Toxin Injection for Treatment of Chronic Anal Fissure: Is There Any Dose-Dependent Efficiency? A Meta-Analysis. World J Surg. 2016 Dec;40(12):3064-3072. doi: 10.1007/s00268-016-3693-9. PMID 27539490
- [Background] Nasr M, Ezzat H, Elsebae M. Botulinum toxin injection versus lateral internal sphincterotomy in the treatment of chronic anal fissure: a randomized controlled trial. World J Surg. 2010 Nov;34(11):2730-4. doi: 10.1007/s00268-010-0736-5. PMID 20703472
- [Background] Valizadeh N, Jalaly NY, Hassanzadeh M, Kamani F, Dadvar Z, Azizi S, Salehimarzijarani B. Botulinum toxin injection versus lateral internal sphincterotomy for the treatment of chronic anal fissure: randomized prospective controlled trial. Langenbecks Arch Surg. 2012 Oct;397(7):1093-8. doi: 10.1007/s00423-012-0948-2. Epub 2012 Mar 20. PMID 22430300
- [Background] Magdy A, El Nakeeb A, Fouda el Y, Youssef M, Farid M. Comparative study of conventional lateral internal sphincterotomy, V-Y anoplasty, and tailored lateral internal sphincterotomy with V-Y anoplasty in the treatment of chronic anal fissure. J Gastrointest Surg. 2012 Oct;16(10):1955-62. doi: 10.1007/s11605-012-1984-5. Epub 2012 Aug 7. PMID 22869534
- [Background] Katsinelos P, Papaziogas B, Koutelidakis I, Paroutoglou G, Dimiropoulos S, Souparis A, Atmatzidis K. Topical 0.5% nifedipine vs. lateral internal sphincterotomy for the treatment of chronic anal fissure: long-term follow-up. Int J Colorectal Dis. 2006 Mar;21(2):179-83. doi: 10.1007/s00384-005-0766-x. Epub 2005 Aug 10. PMID 16091912
- [Background] Chen HL, Woo XB, Wang HS, Lin YJ, Luo HX, Chen YH, Chen CQ, Peng JS. Botulinum toxin injection versus lateral internal sphincterotomy for chronic anal fissure: a meta-analysis of randomized control trials. Tech Coloproctol. 2014 Aug;18(8):693-8. doi: 10.1007/s10151-014-1121-4. Epub 2014 Feb 6. PMID 24500725
- [Background] Bagrasaryan LS, Surgical treatment of anal fissure with anal sphincter pneumodivulsion. 2010: p. 115
- [Background] Delechenaut P, Leroi AM, Weber J, Touchais JY, Czernichow P, Denis P. Relationship between clinical symptoms of anal incontinence and the results of anorectal manometry. Dis Colon Rectum. 1992 Sep;35(9):847-9. doi: 10.1007/BF02047871. PMID 1511644
- [Background] Hyman N. Incontinence after lateral internal sphincterotomy: a prospective study and quality of life assessment. Dis Colon Rectum. 2004 Jan;47(1):35-8. doi: 10.1007/s10350-003-0002-0. Epub 2004 Jan 14. PMID 14719148
- [Background] Sultan AH, Kamm MA, Hudson CN, Thomas JM, Bartram CI. Anal-sphincter disruption during vaginal delivery. N Engl J Med. 1993 Dec 23;329(26):1905-11. doi: 10.1056/NEJM199312233292601. PMID 8247054
- [Background] Tjandra JJ, Han WR, Ooi BS, Nagesh A, Thorne M. Faecal incontinence after lateral internal sphincterotomy is often associated with coexisting occult sphincter defects: a study using endoanal ultrasonography. ANZ J Surg. 2001 Oct;71(10):598-602. doi: 10.1046/j.1445-2197.2001.02211.x. PMID 11552935
- [Background] Zetterstrom J, Mellgren A, Jensen LL, Wong WD, Kim DG, Lowry AC, Madoff RD, Congilosi SM. Effect of delivery on anal sphincter morphology and function. Dis Colon Rectum. 1999 Oct;42(10):1253-60. doi: 10.1007/BF02234209. PMID 10528760
- [Background] Khubchandani IT, Reed JF. Sequelae of internal sphincterotomy for chronic fissure in ano. Br J Surg. 1989 May;76(5):431-4. doi: 10.1002/bjs.1800760504. PMID 2736353
- [Background] Zbar A., M. Aslam, and V. Allgar, Faecal incontinence after internal sphincterotomy for anal fissure. Techniques in Coloproctology, 2000. 4(1): p. 25-28.
- [Background] Zharkov, EE, Comprehensive treatment of chronic anal fissure. 2009: p. 126.
- [Background] Iswariah H, Stephens J, Rieger N, Rodda D, Hewett P. Randomized prospective controlled trial of lateral internal sphincterotomy versus injection of botulinum toxin for the treatment of idiopathic fissure in ano. ANZ J Surg. 2005 Jul;75(7):553-5. doi: 10.1111/j.1445-2197.2005.03427.x. PMID 15972045
- [Background] Nelson RL, Thomas K, Morgan J, Jones A. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003431. doi: 10.1002/14651858.CD003431.pub3. PMID 22336789
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Jorge JM, Wexner SD. Anorectal manometry: techniques and clinical applications. South Med J. 1993 Aug;86(8):924-31. doi: 10.1097/00007611-199308000-00016. PMID 8351556